CLINICAL TRIAL: NCT04004988
Title: A Study to Compare the Pharmacokinetics of Tirzepatide Administered Subcutaneously by an Autoinjector Versus Prefilled Syringe in Healthy Subjects
Brief Title: A Study of Tirzepatide Administered by Two Different Devices in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17105; I8F-MC-GPGS (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide Test (Experimental): Participants received single dose of 5 milligram (mg) Tirzepatide by subcutaneous injection (SC) via an autoinjector (AI) in one of two study periods.
  Interventions: Drug: Tirzepatide; Device: Auto-injector (AI)
- Tirzepatide Reference (Experimental): Participants received single dose of 5mg Tirzepatide by subcutaneous injection (SC) via a prefilled syringe (PFS) in one of two study periods.
  Interventions: Drug: Tirzepatide; Device: Prefilled syringe (PFS)

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
Device: Prefilled syringe (PFS) — PFS used to administer tirzepatide
  Arms: Tirzepatide Reference
Device: Auto-injector (AI) — AI used to administer tirzepatide
  Arms: Tirzepatide Test

SUMMARY:
The purpose of this study is to compare the amount of tirzepatide that gets into the blood stream and how long it takes the body to get rid of it, when given as a solution formulation via an autoinjector versus a conventional prefilled syringe. The tolerability of tirzepatide will also be evaluated and information about any adverse effects experienced will be collected.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be about 14 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of nonchildbearing potential as determined by medical history, physical examination, and other screening procedures
* Are between the body mass index (BMI) of 18.0 and 32.0 kilograms per meter squared (kg/m²), inclusive, at screening
* Are agreeable to receiving study treatment by injections under the skin

Exclusion Criteria:

* Have known allergies to tirzepatide or related compounds
* Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase or GI disorder (eg, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors
* Have a prior history of malignant disease(s) in the past 5 years prior to screening
* Smoke more than the equivalent of 10 cigarettes per day
* Is a known user of drugs of abuse

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Nus Centre for Clin Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: Participants received single dose of 5 milligram (mg) tirzepatide by subcutaneous injection (SC) administered through autoinjector on day 1 of period 1.
  Participants received single dose of 5 mg tirzepatide by SC injection administered through prefilled syringe on day 1 of period 2.
- Sequence B: Participants received single dose of 5 mg tirzepatide by SC injection administered through prefilled syringe on day 1 of period 1.
  Participants received single dose of 5 mg tirzepatide by SC injection administered through autoinjector on day 1 of period 2.
Period: Period 1
Arm/Group | Sequence A | Sequence B
Started | 24 | 23
Received at Least One Dose of Study Drug | 22 | 23
Completed | 21 | 20
Not Completed | 3 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 2
Period: Period 2
Arm/Group | Sequence A | Sequence B
Started | 21 | 20
Received at Least One Dose of Study Drug | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- All Participants: Participants received 5mg of tirzepatide by SC injection administered by autoinjector or prefilled syringe on day 1 of each period as per the dosing sequence.
Arm/Group | All Participants
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 47
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 47

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide From Time Zero to Infinity (AUC0toinf)
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Tirzepatide from Time Zero to Infinity (AUC0toinf) was reported.
Time Frame: Predose, 8hours(h), 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 168h, 336h , 480h, 864h postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*h/mL)
Groups:
- 5 mg Tirzepatide AI: Participants received single dose of 5 mg tirzepatide by SC injection administered through autoinjector.
- 5 mg Tirzepatide PFS: Participants received single dose of 5mg tirzepatide by SC injection administered through prefilled syringe.
Arm/Group | 5 mg Tirzepatide AI | 5 mg Tirzepatide PFS
Number analyzed (Participants) | 42 | 42
Nanogram*hour per milliliter (ng*h/mL) | 101000 (18) | 104000 (18)

2. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Tirzepatide
Description: PK: Maximum Observed Plasma Concentration (Cmax) of Tirzepatide was reported
Time Frame: Predose, 8hours(h), 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 168h, 336h , 480h, 864h postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Milliliter (ng/mL)
Groups:
- 5 mg Tirzepatide PFS: Participants received single dose of 5 mg tirzepatide by SC injection administered through prefilled syringe.
Arm/Group | 5 mg Tirzepatide AI | 5 mg Tirzepatide PFS
Number analyzed (Participants) | 42 | 44
Nanogram per Milliliter (ng/mL) | 530 (25) | 556 (22)

ADVERSE EVENTS:
Time Frame: Up to 72 days
Description: All participants who received at least one dose of study drug.
Arm/Group | 5 mg Tirzepatide AI | 5 mg Tirzepatide PFS
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/44
Other Adverse Events (participants affected / at risk) | 40/42 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide AI (N=42) | 5 mg Tirzepatide PFS (N=44)
Catheter site phlebitis (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide AI (N=42) | 5 mg Tirzepatide PFS (N=44)
Abdominal distension (Gastrointestinal disorders) | 20 (21) | 29 (34)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Eructation (Gastrointestinal disorders) | 5 (6) | 8 (8)
Nausea (Gastrointestinal disorders) | 14 (14) | 12 (13)
Vomiting (Gastrointestinal disorders) | 14 (26) | 16 (31)
Catheter site bruise (General disorders) | 3 (4) | 6 (6)
Catheter site erythema (General disorders) | 4 (5) | 6 (6)
Catheter site phlebitis (General disorders) | 0 (0) | 3 (3)
Catheter site swelling (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 0 (0) | 3 (3)
Vessel puncture site bruise (General disorders) | 7 (8) | 2 (2)
Vessel puncture site phlebitis (General disorders) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 24 (24) | 22 (22)
Dizziness (Nervous system disorders) | 3 (4) | 2 (3)
Headache (Nervous system disorders) | 8 (11) | 11 (12)
Lethargy (Nervous system disorders) | 3 (3) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT04004988/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT04004988/SAP_001.pdf